CLINICAL TRIAL: NCT05170854
Title: The Impact of Liver Cirrhosis on Outcomes in Trauma Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 042.HEP.2018.D
Record Dates: First submitted 2019-08-12; First posted 2021-12-28 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Cirrhosis
Keywords: cirrhotic trauma
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Given that there are only a few studies on the effects of cirrhosis on trauma patients and none have addressed the impact cirrhosis has on the incidence of infections, it is important that we study this to determine the mortality in cirrhotic trauma patients and ascertain the incidence of infectious complications in these patients. We hypothesize that trauma patients with cirrhosis will have higher rates of mortality and infectious complications.

DETAILED DESCRIPTION:
There have been a select few studies addressing the effects of cirrhosis on trauma patients. These studies show an increase in morbidity and mortality. However, there is limitation in the depth and breadth of analysis. The primary aim of this study is to determine the mortality rates in cirrhotic trauma patients with a secondary end-point being the determination of the incidence of infections associated with these patients.

Given that there are only a few studies on the effects of cirrhosis on trauma patients and none have addressed the impact cirrhosis has on the incidence of infections, it is important that we study this to determine the mortality in cirrhotic trauma patients and ascertain the incidence of infectious complications in these patients. PI hypothesizes that trauma patients with cirrhosis will have higher rates of mortality and infectious complications.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic trauma patients in the United States within 2010-2018
* Patients ≥ 18 years old

Exclusion Criteria:

* Patients less than 18 years old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed diagnosis of cirrhosis via radiologic, laboratory profile and intraoperative findings will be selected.Data will be extracted from the NTDB & TQIP databanks from 2010-2018.
Sampling Method: Non-Probability Sample
Enrollment: 4774035 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Mortality | 2010-2018
  Patient death
Incidence of infectious complications | 2010-2018
  Incidents of complications with infections

SECONDARY OUTCOMES:
Patient demographics | 2010-2018
  demographics of patients
vital signs; clinical measurements | 2010-2018
  clinical measurements
vital signs; pulse rate | 2010-2018
  pulse rate (bpm)
vital signs; temperature | 2010-2018
  temperature
vital signs; respiration rate | 2010-2018
  respiration rate
vital signs; blood pressure | 2010-2018
  blood pressure
injury characteristics | 2010-2018
  characteristics of injuries
hospital and ICU lengths of stay | 2010-2018
  length of days patients stays in hospital/ICU
transfusion data | 2010-2018
  data regarding transfusions
alcohol use indicator | 2010-2018
  indicator of alcohol use
drug use indicator | 2010-2018
  indicator of drug use
ventilator days | 2010-2018
  days on ventilator
Abbreviated Injury Scale | 2010-2018
  abbreviated injury scale score
Glasgow Coma Scale | 2010-2018
  glasgow coma scale score
Injury Severity Score | 2010-2018
  score of injury
discharge date | 2010-2018
  date of discharge
arrival date | 2010-2018
  date of arrival

CONTACTS AND LOCATIONS:
Overall Officials: Parvez Mantry, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Health System, Dallas, Texas, United States